CLINICAL TRIAL: NCT03229577
Title: Yale Wellness Project Randomized Controlled Trial
Brief Title: Yale Wellness Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2000020302
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Mental Health Wellness 1
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sudarshan Kriya Yoga (Experimental): Sudarshan Kriya Yoga workshop is a nationally-recognized program focused on teaching yoga-based breathing techniques.
  Interventions: Behavioral: Sudarshan Kriya Yoga
- Mindfulness-Based Stress Reduction (Experimental): Mindfulness-Based Stress Reduction (MBSR) is a nationally-recognized program focused on teaching mindfulness techniques.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Emotional Intelligence (Experimental): Emotional Intelligence is a program developed for university students that focuses on teaching the skills of emotional intelligence such as labeling, understanding, and regulating emotions.
  Interventions: Behavioral: Emotional Intelligence
- Control (No Intervention): The control group will receive no intervention.

INTERVENTIONS:
Behavioral: Sudarshan Kriya Yoga — Yoga-based breathing program.
  Arms: Sudarshan Kriya Yoga
Behavioral: Mindfulness-Based Stress Reduction — Mindfulness program.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Emotional Intelligence — Emotional Intelligence program.
  Other Names: EI
  Arms: Emotional Intelligence

SUMMARY:
The Yale College Emotional Intelligence project aims to highlight the beneficial impact of wellness programs for Yale students. The investigators will examine the benefits of 3 empirically-validated programs (Emotional Intelligence, Mindfulness-Based Stress Reduction (MBSR) & SKY Yoga Breathing) for Yale students on measures of general well-being (e.g. perceived stress, gratitude etc). The study will also include a no-treatment control group as a comparative measure to the well-being programs. The goal of the study is to show how each program benefits student well-being over time. Pre-intervention and post-intervention data will be collected. The hypothesis is that all 3 workshops will decrease stress and improve well-being and that the manner in which each workshop will do so may be different (e.g. MBSR will benefit student well-being by increasing mindfulness and self-compassion whereas Emotional Intelligence may benefit student well-being by improving cognitive emotion regulation). Given the current state of mental health challenges and stress on college campuses, the goal of this randomized-controlled trial is to strengthen the literature on wellness programs for students and to show that student well-being can significantly increase through effective interventions.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Yale student.

Exclusion Criteria:

* Under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Mood and Anxiety Symptom Questionnaire Short Form | 11 Weeks
  The MASQ-Short contains 30 questions with three subscales that measure: general distress, depressive symptoms, and anxious symptoms. All individual items are rated on a scale 1 to 5, where 1 indicates the individual has not felt this way at all during the past week and 5 indicates that they have felt this way extremely. The total possible score for the scale is 150 and the minimum is 30. The three sub scales are totaled together to create the total score (each contains 10 questions). The minimum and maximum scores for the subscales are 10 and 50 respectively.
Perceived Stress Scale | 11 Weeks
  The 10-item Perceived Stress Scale (Cohen, S., Kamarck, T., and Mermelstein, R., 1983) measures the degree to which situations in one's life are appraised as stressful. Respondents report how frequently they feel stress or have difficulty coping with life stresses. Items include questions that ask about the frequency of negative experiences, e.g., "In the last month, how often have you felt that you were unable to control the important things in your life?" and positive experiences, e.g., "In the last month, how often have you felt that things were going your way?" Responses range from 0=never to 4=very often. The minimum and maximum scores are 0 and 40 respectively.
Emotional Intelligence Perception Skill Test | 11 weeks
  Assesses participant ability to perceive emotions accurately
Satisfaction with Life Scale | 11 Weeks
  The Satisfaction with Life Scale (SWLS; Diener, Emmons, Larsen, & Griffin, 1985) will be used to test participants satisfaction with their lives. This scale is 5-items and is rated on a 7 point scale from 1 (strongly disagree) to 7 (strongly agree). Examples of items include, "The conditions of my life are excellent" and " If I could live my life over, I would change almost nothing". The minimum and maximum total scores are 5 and 35 respectively.
Five Facet Mindfulness Questionnaire | 11 Weeks
  Five Facet Mindfulness Questionnaire - 15-item, (FFMQ-15; Baer et al., 2008) is a 15 item measure of mindfulness that participants rate on a scale from 1 - 5 depending on how much they agree with the statement. Low scores indicate low mindfulness and high scores indicate high levels of mindfulness. Minimum and maximum scores are 15 and 75 respectively.
Ryff Scales for Psychological Wellbeing | 11 Weeks
  Psychological Well-Being Scale-18 (Ryff, 2008) is an 18-item form to assess psychological wellbeing. Items are rated on a 7-point scale from strongly disagree to strongly agree. Low scores indicate poor psychological wellbeing while high scores indicate healthy psychological wellbeing. Total scores range from 18 to 126.
Burnout | 11 Weeks
  The Single-item Measure of Burnout (Rohland, Kruse, & Rohrer, 2004) will be used to measure student burnout. This measure only contains one item: "Overall, based on your definition of burnout, how would you rate your level of burnout?" Participants are asked to choose one answer ranging from 1 (I enjoy my work. I have no symptoms of burnout) to 5 (I feel completely burned out and often wonder if I can go on. I am at the point where I may need some changes or may need to seek some sort of help).

SECONDARY OUTCOMES:
Gratitude Scale | 11 Weeks
  The Gratitude Questionnaire-Six Item Form (GQ-6; McCullough, Emmons, & Tsang, 2002) is a 6-item measure to test a participant amount of gratitude that they feel. The items are rated on a scale from 1 to 7, 1 (strongly disagree) to 7 (strongly agree). Examples of items include, "I have so much in my life to be thankful for" and "Long amounts of time can go by before I feel grateful to something or someone." Low scores indicate low gratitude and high scores indicate high gratitude. Total scores range from 6 to 42.
Self-compassion Scale | 11 Weeks
  The 12 item Self-Compassion-Short Form assess self-reported self-compassion. Responses are given on a five-point scale from "Almost Never" to "Almost Always." Low scores indicate low self-compassion and high scores indicate high self-compassion. Scores range from 12 to 60.
Life Orientation Scale | 11 Weeks
  The Life Orientation Test- Revised (LOT-R; Scheier, Carver, & Bridges, 1994) will be used to measure the optimism of students. This test includes 10 items rated on a 5 point scale from 1 ( I disagree a lot) to 5 (I agree a lot). Examples of items include, " If something can go wrong for me, it will" and "In uncertain times, I usually expect the best." Scores range from low optimism (10) to high optimism (50).
Brief COPE Scale | 11 Weeks
  Brief COPE (Carver, 1997) is a 28-item survey for measuring what emotion regulation strategies people use to deal with stressful situations. Participatns are asked to answer questions on a scale from 1 - 4. Low scores of emotion regulation ability (28) to high scores of emotion regulation ability (112).
Creativity Performance Questions | 11 Weeks
  Assesses creativity using performance metrics. Students are asked to come up with as many creative solutions to a prompt over the course of 1.5 minutes. Responses are coded for uniqueness and breadth.
Social Connectedness Scale | 11 Weeks
  This scale consists of 10 positively worded and 10 negatively worded items. The 10 new positively worded items capture experiencing a sense of closeness with others and maintaining and seeking connections. Sample items include "I am able to connect with other people," and "I am able to relate to my peers." The 10 negatively worded items capture one's experience of distance and isolation from others, for example, "I see myself as a loner" and "I feel like an outsider." Items are rated on a 6-point Likert-type scale ranging from "Strongly disagree" to "Strongly agree." Low scores (20) indicate low social connectedness while high scores (80) indicate high school connectedness.
One-item Self-esteem Scale | 11 Weeks
  Single Item Self-Esteem Scale (SISE; Robins, Hendin, & Trzesniewski, 2001) is a single item measure of the construct of self-esteem that has been validated against the well-known Rosenberg Self-Esteem Scale. Scores range from 1 - 5 with low self-esteem indicated by a score of 1.
Big Five Questionnaire | Baseline
  The Big Five Inventory is a 44 item self-report measure for assessing the basic personality dimensions of extraversion (e.g., "talkative"), agreeableness (e.g., "helpful and unselfish with others"), conscientiousness ("does things carefully and completely"), neuroticism, and openness to experience (e.g., "original, comes up with new ideas"; Soto, John, Gosling, & Potter, 2008). Respondents rate the extent to which they agree with self-descriptive statements using a 1 ("strongly disagree") to 5 ("strongly agree") response scale. A total score is not created for this measure. Rather, sub scale scores are created. Ranges of scores: extraversion (8-40), agreeableness (9-45), conscientiousness (9-45), neuroticism (8-40), and openness (10-50).
Human Wellbeing Scale | 11 Weeks
  This scale is a 36-item scale where participants report how often they feel a specific list of emotions. Low scores indicate low wellbeing and high scores indicate high wellbeing. Choices range from 1-5 and scores range from 36 to 180.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Brackett, Ph.D., Principal Investigator — Director, Yale Center for Emotional Intelligence; Leilah Harouni, B.S., Study Chair — Postgraduate Research Associate, Yale Center for Emotional Intelligence
Locations (1):
- Yale Center for Emotional Intelligence, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No